CLINICAL TRIAL: NCT01923467
Title: Project Quit: Positive vs. Negative Offers of an Online Stop Smoking Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Lawrence C. An, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P50CA101451 (NIH)
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2014-12

CONDITIONS: Smoking Cessation
Keywords: smoking; nicotine replacement; internet
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Project Quit plus NRT patches (Experimental): All participants in the program will be offered the opportunity to complete the Project Quit stop smoking program. Project Quit is an individually-tailored, web-based program which has been scientifically proven to help people succeed at their quit attempts. All eligible participants will also receive a 2-week supply of Nicotine patches 21 mg.
  Interventions: Behavioral: Project Quit stop smoking program; Drug: Nicotine patches 21 mg

INTERVENTIONS:
Behavioral: Project Quit stop smoking program — This online stop-smoking program is individually tailored to the participant's readiness to quit, smoking triggers, and many other characteristics. It has been scientifically proven to improve quit success.
Drug: Nicotine patches 21 mg — Eligible participants will receive a 2-week supply of Nicoderm CQ Step 1 patches to help them be successful in their quit attempt.
  Other Names: Nicoderm CQ Step 1 (21 mg)

SUMMARY:
This project is designed to test the effects of affirmation and positive/negative imagery on individuals' thoughts about quitting smoking and willingness to join a stop smoking program. Previous studies have noted that viewing negative images elicits a stronger emotional response, and many stop-smoking campaigns have used such images to push people to quit smoking. However, research also shows that people are generally resistant to health messages. Using affirmation can help to lessen that resistance.

In this study, we use a 2x3 design to study the individual effects of negative imagery and affirmation on smokers' intentions to quit smoking, acceptance of an offer to join a quit smoking program, and program participation and outcomes. We hope to find out whether there is an additive effect of the negative imagery and affirmation on the outcomes listed above. Our specific aims are:

Aim 1: Determine if affirmation increases the uptake of an offer of joining a stop smoking program.

Aim 2: Determine if image type (positive vs. neutral vs. negative) increases the uptake of the stop smoking program offer.

Aim 3: Determine whether there is an interaction between image type and affirmation in people's willingness to join a stop smoking program.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker

Exclusion Criteria:

* Current participation in another stop-smoking program
* Current use of stop smoking medications
* Pregnant or breastfeeding
* Limited internet or email access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C An, MD, Principal Investigator — University of Michigan
Locations (1):
- Center for Health Communications Research, University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Project Quit Plus NRT Patches
Started | 767 (Offered stop smoking program)
Baseline Completed, Enrolled | 288
Completed | 226 (Completed 3-month follow up survey)
Not Completed | 541
Not completed — Lost to Follow-up | 62
Not completed — Subject non-interest | 479

BASELINE CHARACTERISTICS:
Population: Smoker recruited from an online survey panel.
Arm/Group | Project Quit Plus NRT Patches
Number analyzed (Participants) | 767
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398
  Male | 369
Region of Enrollment [Number; unit: participants]
  United States | 767
Number of cigarettes smoked per day [Mean (Standard Deviation); unit: Cigarettes] | 16.0 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Acceptance of Offer to Join Stop Smoking Program
Description: After participation in online image viewing and writing reflection tasks, participants will be asked if they would like to take part in an online stop-smoking program.
Time Frame: 1 Day of Enrollment
Measure: Number; unit: participants
Arm/Group | Project Quit Plus NRT Patches
Number analyzed (Participants) | 767
participants | 288

ADVERSE EVENTS:
Arm/Group | Project Quit Plus NRT Patches
Serious Adverse Events (participants affected / at risk) | 0/767
Other Adverse Events (participants affected / at risk) | 0/767

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No